CLINICAL TRIAL: NCT05812573
Title: A Retrospective Study for Multiple Endocrine Neoplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202302051RINC
Record Dates: First submitted 2023-03-15; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Multiple Endocrine Neoplasia
MeSH Terms: conditions — Multiple Endocrine Neoplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- multiple endocrine neoplasia: patients with multiple endocrine neoplasia
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention, only observation

SUMMARY:
Retrospectively review the clinical characteristics of patients with multiple endocrine neoplasia type I in National Taiwan University Hospital.

DETAILED DESCRIPTION:
The investigators will retrospectively review the clinical characteristics of patients with multiple endocrine neoplasia type I in National Taiwan University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple endocrine neoplasia

Exclusion Criteria:

* Patients younger than 18 years old

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple endocrine neoplasia who age 18 to 99 years old
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2024-02-14 (Estimated)

PRIMARY OUTCOMES:
Number or endocrine organs involved | 2023/2/14-2033/2/14
  The number of endocrine organs involved in MEN patients

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan